CLINICAL TRIAL: NCT02822794
Title: A Phase 3, Multicenter, Randomized, Open-Label Study to Investigate the Efficacy and Safety of Sofosbuvir/Velpatasvir Fixed-Dose Combination and Ribavirin for 12 or 24 Weeks in Subjects With Chronic Genotype 1 or 2 HCV Infection Who Have Previously Failed a Direct-Acting Antiviral-Containing Regimen
Brief Title: Sofosbuvir/Velpatasvir Fixed-Dose Combination and Ribavirin for 12 or 24 Weeks in Participants With Chronic Genotype 1 or 2 Hepatitis C Virus Infection Who Have Previously Failed a Direct-Acting Antiviral-Containing Regimen
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GS-US-342-3921
Record Dates: First submitted 2016-06-30; First posted 2016-07-04 (Estimated); Results first posted 2018-07-03 (Actual); Last update posted 2018-11-14 (Actual); Status verified 2018-07

CONDITIONS: Hepatitis C Virus Infection
MeSH Terms: conditions — Hepatitis C | interventions — sofosbuvir-velpatasvir drug combination; Ribavirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- SOF/VEL FDC + RBV 12 weeks (Experimental): SOF/VEL FDC + RBV for 12 weeks in participants with genotype 1 or 2 HCV infection
  Interventions: Drug: SOF/VEL; Drug: RBV
- SOF/VEL FDC + RBV 24 weeks (Experimental): SOF/VEL FDC + RBV for 24 weeks in participants with genotype 1 or 2 HCV infection
  Interventions: Drug: SOF/VEL; Drug: RBV

INTERVENTIONS:
Drug: SOF/VEL — 400/100 mg tablet administered orally once daily
  Other Names: GS-7977/GS-5816; Epclusa®
Drug: RBV — Capsules administered orally in a divided daily dose according to package insert weight-based dosing recommendations (≤ 60 kg = 600 mg, > 60 kg to ≤ 80 kg = 800 mg, and ≥ 80 kg = 1000 mg)
  Other Names: REBETOL®

SUMMARY:
The primary objective of this study is to evaluate the antiviral efficacy, safety, and tolerability of therapy with sofosbuvir/velpatasvir (SOF/VEL) fixed-dose combination (FDC) and ribavirin (RBV) in participants with chronic genotype 1 or 2 hepatitis C virus (HCV) infection who have previously failed a direct-acting antiviral (DAA)-containing regimen.

ELIGIBILITY:
Key Inclusion Criteria:

* Genotype 1 or 2 HCV infection
* Chronic HCV infection (≥ 6 months prior to screening) documented by prior medical history or liver biopsy
* Previously treated with a DAA-containing regimen of at least 4 week duration

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 117 (Actual)
Dates: Start 2016-07-25 (Actual); Primary Completion 2017-06-02 (Actual); Study Completion 2017-08-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (18):
- Japan (18):
  - Ehime
  - Hiroshima
  - Ichikawa-shi
  - Iruma-gun
  - Kashihara
  - Kurume-shi
  - Kyoto
  - Maebashi
  - Musashino-shi
  - Nagoya
  - Nishinomiya
  - Okayama
  - Ōgaki
  - Ōmura
  - Sapporo
  - Suita
  - Takamatsu
  - Yamagata

IPD SHARING:
Plan to Share IPD: Yes
Qualified external researchers may request IPD for this study after study completion. For more information, please visit our website at http://www.gilead.com/research/disclosure-and-transparency.
Supporting Information: Study Protocol, SAP
Time Frame: 18 months after study completion
Access Criteria: A secured external environment with username, password, and RSA code.
URL: http://www.gilead.com/research/disclosure-and-transparency

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study sites in Japan. The first participant was screened on 25 July 2016. The last study visit occurred on 25 August 2017.
Pre-assignment Details: 132 participants were screened.
Groups:
- SOF/VEL FDC + RBV 12 Weeks: Sofosbuvir/velpatasvir (SOF/VEL) (400/100 mg) fixed-dose combination (FDC) tablet orally once daily + ribavirin (RBV) capsule (600, 800, or 1000 mg daily based on weight) for 12 weeks
- SOF/VEL FDC + RBV 24 Weeks: SOF/VEL (400/100 mg) FDC tablet orally once daily + RBV capsule (600, 800, or 1000 mg daily based on weight) for 24 weeks
Period: Overall Study
Arm/Group | SOF/VEL FDC + RBV 12 Weeks | SOF/VEL FDC + RBV 24 Weeks
Started | 57 | 60
Completed | 56 | 60
Not Completed | 1 | 0
Not completed — Withdrew Consent | 1 | 0

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set: participants who received at least 1 dose of study drug
Groups:
- SOF/VEL+RBV 12 Weeks (GT1): SOF/VEL (400/100 mg) FDC tablet orally once daily + RBV capsule (600, 800, or 1000 mg daily based on weight) for 12 weeks in participants with genotype 1 (GT1) HCV infection
- SOF/VEL+RBV 12 Weeks (GT2): SOF/VEL (400/100 mg) FDC tablet orally once daily + RBV capsule (600, 800, or 1000 mg daily based on weight) for 12 weeks in participants with genotype 2 (GT2) HCV infection
- SOF/VEL+RBV 24 Weeks (GT1): SOF/VEL (400/100 mg) FDC tablet orally once daily + RBV capsule (600, 800, or 1000 mg daily based on weight) for 24 weeks in participants with genotype 1 (GT1) HCV infection
- SOF/VEL+RBV 24 Weeks (GT2): SOF/VEL (400/100 mg) FDC tablet orally once daily + RBV capsule (600, 800, or 1000 mg daily based on weight) for 24 weeks in participants with genotype 2 (GT2) HCV infection
- Total: Total of all reporting groups
Arm/Group | SOF/VEL+RBV 12 Weeks (GT1) | SOF/VEL+RBV 12 Weeks (GT2) | SOF/VEL+RBV 24 Weeks (GT1) | SOF/VEL+RBV 24 Weeks (GT2) | Total
Number analyzed (Participants) | 47 | 10 | 48 | 12 | 117
Age, Continuous [Mean (Standard Deviation); unit: years] | 63 (9.7) | 59 (15.7) | 64 (10.1) | 61 (7.2) | 63 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 5 | 28 | 5 | 67
  Male | 18 | 5 | 20 | 7 | 50
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 47 | 10 | 48 | 12 | 117
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Not Hispanic or Latino | 47 | 10 | 48 | 12 | 117
HCV genotype [Count of Participants; unit: Participants]
  Genotype 1a | 2 | 0 | 1 | 0 | 3
  Genotype 1b | 45 | 0 | 47 | 0 | 92
  Genotype 2a/2c | 0 | 3 | 0 | 4 | 7
  Genotype 2b | 0 | 2 | 0 | 4 | 6
  Genotype 2 (No Confirmed Subtype) | 0 | 5 | 0 | 4 | 9
IL28b Status [Count of Participants; unit: Participants] — The CC, CT, and TT alleles are different forms of the IL28b gene.
  Participants
    CC | 15 | 8 | 21 | 6 | 50
    CT | 28 | 1 | 20 | 6 | 55
    TT | 4 | 1 | 7 | 0 | 12
HCV RNA (log10 IU/mL) [Mean (Standard Deviation); unit: log10 IU/mL] | 6.2 (.47) | 6.6 (.46) | 6.2 (.51) | 6.2 (.86) | 6.2 (.54)
HCV RNA Category [Count of Participants; unit: Participants]
  < 800,000 IU/mL | 10 | 1 | 10 | 4 | 25
  ≥ 800,000 IU/mL | 37 | 9 | 38 | 8 | 92

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Sustained Virologic Response (SVR) 12 Weeks After Discontinuation of Therapy (SVR12)
Description: SVR12 was defined as HCV RNA < the lower limit of quantitation (LLOQ; ie, 15 IU/mL) at 12 weeks after stopping study treatment.
Time Frame: Posttreatment Week 12
Population: Full Analysis Set: participants who were randomized and received at least 1 dose of study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | SOF/VEL+RBV 12 Weeks (GT1) | SOF/VEL+RBV 12 Weeks (GT2) | SOF/VEL+RBV 24 Weeks (GT1) | SOF/VEL+RBV 24 Weeks (GT2)
Number analyzed (Participants) | 47 | 10 | 48 | 12
percentage of participants | 85.1 [71.7 to 93.8] | 70.0 [34.8 to 93.3] | 97.9 [88.9 to 99.9] | 91.7 [61.5 to 99.8]
Statistical Analysis 1: Comparison: SOF/VEL+RBV 12 Weeks (GT1); Test type: Superiority; p < 0.001, Binomial test; P-value is obtained from the 2-sided exact 1-sample binomial test for the superiority of SOF/VEL+RBV 12 Weeks (GT1) over the performance goal of 50%
Statistical Analysis 2: Comparison: SOF/VEL+RBV 24 Weeks (GT1); Test type: Superiority; p < 0.001, Binomial test; P-value is obtained from the 2-sided exact 1-sample binomial test for the superiority of SOF/VEL +RBV 24 Weeks (GT1) over the performance goal of 50%

2. Primary Outcome: Percentage of Participants Who Permanently Discontinued Any Study Drug Due to an Adverse Event
Time Frame: Up to 24 weeks
Population: Safety Analysis Set
Measure: Number; unit: percentage of participants
Groups:
- SOF/VEL+RBV 12 Weeks: SOF/VEL (400/100 mg) FDC tablet orally once daily + RBV capsule (600, 800, or 1000 mg daily based on weight) for 12 weeks in participants with genotype 1 or 2 HCV infection
- SOF/VEL+RBV 24 Weeks: SOF/VEL (400/100 mg) FDC tablet orally once daily + RBV capsule (600, 800, or 1000 mg daily based on weight) for 24 weeks in participants with genotype 1 or 2 HCV infection
Arm/Group | SOF/VEL+RBV 12 Weeks | SOF/VEL+RBV 24 Weeks
Number analyzed (Participants) | 57 | 60
percentage of participants | 1.8 | 3.3

3. Secondary Outcome: Percentage of Participants With SVR at 4 Weeks After Discontinuation of Therapy (SVR4)
Description: SVR4 was defined as HCV RNA < LLOQ at 4 weeks after stopping study treatment.
Time Frame: Posttreatment Week 4
Population: Full Analysis Set
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- SOF/VEL+RBV 12 Weeks: SOF/VEL (400/100 mg) FDC tablet orally once daily + RBV capsule (600, 800, or 1000 mg daily based on weight) for 12 weeks in participants with genotype 1 or genotype 2 HCV infection
- SOF/VEL+RBV 24 Weeks: SOF/VEL (400/100 mg) FDC tablet orally once daily + RBV capsule (600, 800, or 1000 mg daily based on weight) for 24 weeks in participants with genotype 1 or genotype 2 HCV infection
Arm/Group | SOF/VEL+RBV 12 Weeks | SOF/VEL+RBV 24 Weeks
Number analyzed (Participants) | 57 | 60
percentage of participants | 86.0 [74.2 to 93.7] | 98.3 [91.1 to 100.0]

4. Secondary Outcome: Percentage of Participants With SVR at 24 Weeks After Discontinuation of Therapy (SVR24)
Description: SVR 24 was defined as HCV RNA < LLOQ at 24 weeks after stopping study treatment.
Time Frame: Posttreatment Week 24
Population: Full Analysis Set
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | SOF/VEL+RBV 12 Weeks | SOF/VEL+RBV 24 Weeks
Number analyzed (Participants) | 57 | 60
percentage of participants | 82.5 [70.1 to 91.3] | 96.7 [88.5 to 99.6]

5. Secondary Outcome: Percentage of Participants With HCV RNA < LLOQ at Week 1
Time Frame: Week 1
Population: Full Analysis Set
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | SOF/VEL+RBV 12 Weeks | SOF/VEL+RBV 24 Weeks
Number analyzed (Participants) | 57 | 60
percentage of participants | 21.1 [11.4 to 33.9] | 25.0 [14.7 to 37.9]

6. Secondary Outcome: Percentage of Participants With HCV RNA < LLOQ at Week 2
Time Frame: Week 2
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | SOF/VEL+RBV 12 Weeks | SOF/VEL+RBV 24 Weeks
Number analyzed (Participants) | 56 | 60
percentage of participants | 64.3 [50.4 to 76.6] | 70.0 [56.8 to 81.2]

7. Secondary Outcome: Percentage of Participants With HCV RNA < LLOQ at Week 3
Time Frame: Week 3
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | SOF/VEL+RBV 12 Weeks | SOF/VEL+RBV 24 Weeks
Number analyzed (Participants) | 56 | 60
percentage of participants | 91.1 [80.4 to 97.0] | 90.0 [79.5 to 96.2]

8. Secondary Outcome: Percentage of Participants With HCV RNA < LLOQ at Week 4
Time Frame: Week 4
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | SOF/VEL+RBV 12 Weeks | SOF/VEL+RBV 24 Weeks
Number analyzed (Participants) | 56 | 60
percentage of participants | 98.2 [90.4 to 100.0] | 98.3 [91.1 to 100.0]

9. Secondary Outcome: Percentage of Participants With HCV RNA < LLOQ at Week 5
Time Frame: Week 5
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | SOF/VEL+RBV 12 Weeks | SOF/VEL+RBV 24 Weeks
Number analyzed (Participants) | 56 | 60
percentage of participants | 98.2 [90.4 to 100.0] | 98.3 [91.1 to 100.0]

10. Secondary Outcome: Percentage of Participants With HCV RNA < LLOQ at Week 6
Time Frame: Week 6
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | SOF/VEL+RBV 12 Weeks | SOF/VEL+RBV 24 Weeks
Number analyzed (Participants) | 56 | 60
percentage of participants | 100.0 [93.6 to 100.0] | 98.3 [91.1 to 100.0]

11. Secondary Outcome: Percentage of Participants With HCV RNA < LLOQ at Week 8
Time Frame: Week 8
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | SOF/VEL+RBV 12 Weeks | SOF/VEL+RBV 24 Weeks
Number analyzed (Participants) | 56 | 60
percentage of participants | 100.0 [93.6 to 100.0] | 100.0 [94.0 to 100.0]

12. Secondary Outcome: Percentage of Participants With HCV RNA < LLOQ at Week 10
Time Frame: Week 10
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | SOF/VEL+RBV 12 Weeks | SOF/VEL+RBV 24 Weeks
Number analyzed (Participants) | 56 | 59
percentage of participants | 100.0 [93.6 to 100.0] | 100.0 [93.9 to 100.0]

13. Secondary Outcome: Percentage of Participants With HCV RNA < LLOQ at Week 12
Time Frame: Week 12
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | SOF/VEL+RBV 12 Weeks | SOF/VEL+RBV 24 Weeks
Number analyzed (Participants) | 56 | 59
percentage of participants | 100.0 [93.6 to 100.0] | 100.0 [93.9 to 100.0]

14. Secondary Outcome: Percentage of Participants With HCV RNA < LLOQ at Week 16
Time Frame: Week 16
Population: Participants in the Full Analysis Set from the SOF/VEL+RBV 24 Weeks Group with available data were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | SOF/VEL+RBV 24 Weeks
Number analyzed (Participants) | 58
percentage of participants | 100.0 [93.8 to 100.0]

15. Secondary Outcome: Percentage of Participants With HCV RNA < LLOQ at Week 20
Time Frame: Week 20
Population: Participants in the Full Analysis Set from the SOF/VEL+RBV 24 Weeks Group with available data were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | SOF/VEL+RBV 24 Weeks
Number analyzed (Participants) | 58
percentage of participants | 100.0 [93.8 to 100.0]

16. Secondary Outcome: Percentage of Participants With HCV RNA < LLOQ at Week 24
Time Frame: Week 24
Population: Participants in the Full Analysis Set from the SOF/VEL+RBV 24 Weeks Group with available data were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | SOF/VEL+RBV 24 Weeks
Number analyzed (Participants) | 58
percentage of participants | 100.0 [93.8 to 100.0]

17. Secondary Outcome: Change From Baseline in HCV RNA at Week 1
Time Frame: Baseline; Week 1
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: log10 IU/mL
Arm/Group | SOF/VEL+RBV 12 Weeks | SOF/VEL+RBV 24 Weeks
Number analyzed (Participants) | 57 | 60
log10 IU/mL | -4.40 (0.640) | -4.36 (0.698)

18. Secondary Outcome: Change From Baseline in HCV RNA at Week 2
Time Frame: Baseline; Week 2
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: log10 IU/mL
Arm/Group | SOF/VEL+RBV 12 Weeks | SOF/VEL+RBV 24 Weeks
Number analyzed (Participants) | 56 | 60
log10 IU/mL | -4.91 (0.510) | -4.89 (0.603)

19. Secondary Outcome: Change From Baseline in HCV RNA at Week 3
Time Frame: Baseline; Week 3
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: log10 IU/mL
Arm/Group | SOF/VEL+RBV 12 Weeks | SOF/VEL+RBV 24 Weeks
Number analyzed (Participants) | 56 | 60
log10 IU/mL | -5.07 (0.506) | -5.02 (0.575)

20. Secondary Outcome: Change From Baseline in HCV RNA at Week 4
Time Frame: Baseline; Week 4
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: log10 IU/mL
Arm/Group | SOF/VEL+RBV 12 Weeks | SOF/VEL+RBV 24 Weeks
Number analyzed (Participants) | 56 | 60
log10 IU/mL | -5.12 (0.486) | -5.04 (0.580)

21. Secondary Outcome: Change From Baseline in HCV RNA at Week 5
Time Frame: Baseline; Week 5
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: log10 IU/mL
Arm/Group | SOF/VEL+RBV 12 Weeks | SOF/VEL+RBV 24 Weeks
Number analyzed (Participants) | 56 | 60
log10 IU/mL | -5.13 (0.487) | -5.05 (0.579)

22. Secondary Outcome: Change From Baseline in HCV RNA at Week 6
Time Frame: Baseline; Week 6
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: log10 IU/mL
Arm/Group | SOF/VEL+RBV 12 Weeks | SOF/VEL+RBV 24 Weeks
Number analyzed (Participants) | 56 | 60
log10 IU/mL | -5.13 (0.492) | -5.05 (0.579)

23. Secondary Outcome: Change From Baseline in HCV RNA at Week 8
Time Frame: Baseline; Week 8
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: log10 IU/mL
Arm/Group | SOF/VEL+RBV 12 Weeks | SOF/VEL+RBV 24 Weeks
Number analyzed (Participants) | 56 | 60
log10 IU/mL | -5.13 (0.492) | -5.06 (0.584)

24. Secondary Outcome: Change From Baseline in HCV RNA at Week 10
Time Frame: Baseline; Week 10
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: log10 IU/mL
Arm/Group | SOF/VEL+RBV 12 Weeks | SOF/VEL+RBV 24 Weeks
Number analyzed (Participants) | 56 | 59
log10 IU/mL | -5.13 (0.492) | -5.06 (0.589)

25. Secondary Outcome: Change From Baseline in HCV RNA at Week 12
Time Frame: Baseline; Week 12
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: log10 IU/mL
Arm/Group | SOF/VEL+RBV 12 Weeks | SOF/VEL+RBV 24 Weeks
Number analyzed (Participants) | 56 | 59
log10 IU/mL | -5.13 (0.492) | -5.06 (0.589)

26. Secondary Outcome: Change From Baseline in HCV RNA at Week 16
Time Frame: Baseline; Week 16
Population: Participants in the Full Analysis Set from the SOF/VEL+RBV 24 Weeks Group with available data were analyzed.
Measure: Mean (Standard Deviation); unit: log10 IU/mL
Arm/Group | SOF/VEL+RBV 24 Weeks
Number analyzed (Participants) | 58
log10 IU/mL | -5.06 (0.594)

27. Secondary Outcome: Change From Baseline in HCV RNA at Week 20
Time Frame: Baseline; Week 20
Population: Participants in the Full Analysis Set from the SOF/VEL+RBV 24 Weeks Group with available data were analyzed.
Measure: Mean (Standard Deviation); unit: log10 IU/mL
Arm/Group | SOF/VEL+RBV 24 Weeks
Number analyzed (Participants) | 58
log10 IU/mL | -5.06 (0.594)

28. Secondary Outcome: Change From Baseline in HCV RNA at Week 24
Time Frame: Baseline; Week 24
Population: Participants in the Full Analysis Set from the SOF/VEL+RBV 24 Weeks Group with available data were analyzed.
Measure: Mean (Standard Deviation); unit: log10 IU/mL
Arm/Group | SOF/VEL+RBV 24 Weeks
Number analyzed (Participants) | 58
log10 IU/mL | -5.06 (0.594)

29. Secondary Outcome: Percentage of Participants With Overall Virologic Failure
Description: Virologic failure was defined as:
  * On-treatment virologic failure:
    * Breakthrough (confirmed HCV RNA ≥ LLOQ after having previously had HCV RNA < LLOQ while on treatment), or
    * Rebound (confirmed > 1 log10 IU/mL increase in HCV RNA from nadir while on treatment), or
    * Non-response (HCV RNA persistently ≥ LLOQ through 8 weeks of treatment)
  * Virologic relapse:
    * Confirmed HCV RNA ≥ LLOQ during the posttreatment period having achieved HCV RNA < LLOQ at last on-treatment visit.
Time Frame: Up to Posttreatment Week 24
Population: Full Analysis Set
Measure: Number; unit: percentage of participants
Arm/Group | SOF/VEL+RBV 12 Weeks | SOF/VEL+RBV 24 Weeks
Number analyzed (Participants) | 57 | 60
percentage of participants | 15.8 | 3.3

ADVERSE EVENTS:
Time Frame: Adverse Events and Serious Adverse Events: Up to 24 weeks + 30 days. All-Cause Mortality: Up to Posttreatment Week 24.
Description: Safety Analysis Set: participants who received at least 1 dose of study drug
Arm/Group | SOF/VEL+RBV 12 Weeks | SOF/VEL+RBV 24 Weeks
All-Cause Mortality (participants affected / at risk) | 0/57 | 0/60
Serious Adverse Events (participants affected / at risk) | 0/57 | 4/60
Other Adverse Events (participants affected / at risk) | 43/57 | 38/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SOF/VEL+RBV 12 Weeks (N=57) | SOF/VEL+RBV 24 Weeks (N=60)
Pneumonia (Infections and infestations) | 0 | 1
Hepatic angiosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | SOF/VEL+RBV 12 Weeks (N=57) | SOF/VEL+RBV 24 Weeks (N=60)
Anaemia (Blood and lymphatic system disorders) | 14 | 13
Abdominal pain upper (Gastrointestinal disorders) | 3 | 0
Nausea (Gastrointestinal disorders) | 5 | 1
Stomatitis (Gastrointestinal disorders) | 5 | 3
Malaise (General disorders) | 1 | 3
Gastroenteritis (Infections and infestations) | 0 | 4
Oral herpes (Infections and infestations) | 0 | 3
Pharyngitis (Infections and infestations) | 3 | 3
Viral upper respiratory tract infection (Infections and infestations) | 20 | 13
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 1
Headache (Nervous system disorders) | 11 | 2
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 4
Eczema (Skin and subcutaneous tissue disorders) | 4 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 4
Rash (Skin and subcutaneous tissue disorders) | 2 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years

DOCUMENTS (2):
  • Statistical Analysis Plan (2017-06-13): https://cdn.clinicaltrials.gov/large-docs/94/NCT02822794/SAP_000.pdf
  • Study Protocol (2016-06-13): https://cdn.clinicaltrials.gov/large-docs/94/NCT02822794/Prot_001.pdf